CLINICAL TRIAL: NCT00402636
Title: Prospective, Randomized Trial of Rapamycin Plus Estradiol-Eluting Stents Versus Rapamycin-Eluting Stents For The Reduction of Coronary Restenosis (ISAR-PEACE)
Brief Title: Rapamycin+Estradiol- vs. Rapamycin-Eluting Stents to Reduce Restenosis (ISAR-PEACE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S02505
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): rapamycin plus 17beta estradiolvalerat-eluting stent
  Interventions: Device: rapamycin plus 17beta estradiolvalerat-eluting stent
- 2 (Experimental): rapamycin-eluting stent
  Interventions: Device: rapamycin-eluting stent

INTERVENTIONS:
Device: rapamycin plus 17beta estradiolvalerat-eluting stent — rapamycin plus 17beta estradiolvalerat-eluting stent was implanted due to randomisation
  Arms: 1
Device: rapamycin-eluting stent — rapamycin-eluting stent was implanted due to randomisation
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate whether adding estradiol to rapamycin better prevents coronary artery reblockage after drug-eluting stent implantation.

DETAILED DESCRIPTION:
Coronary artery reblockage remains still a drawback of percutaneous coronary interventions even in the era of drug-eluting stents (DES). DESs working principle consists of the delivery of controlled amounts of antiproliferative agents at the local level, which results in the suppression of neontimal proliferation, the main cause of lumen re-narrowing after stent implantation. At present, several DES platforms have been developed and evaluated for clinical use. They differ between them with regard to the stent type, anti-proliferative drug, presence or absence of polymers employed for drug storage and modification of drug-release kinetics as well as type of polymer used for this purpose. Although their mid-term efficacy has been well-established, there is an ongoing debate on the potential of an increased incidence of late stent thrombosis, particularly after discontinuation of thienopyridine therapy, as well as of delayed onset of restenosis or catch-up phenomenon with DESs. Based on animal and human pathological data, investigators have linked the above-mentioned concerns to the presence of permanent polymers in DESs, which have a proinflammatory and prothrombogenic potential, and sometimes may induce a hypersensitivity reaction. On the other hand, lack of or delayed reendothelialization is considered an important factor for development of coronary reblockage. Estradiol has been shown to promote rapid reendothelialization of the stent and to reduce the restenosis after PCI. This trial will compare the anti-restenotic efficacy of the polymer-free rapamycin plus 17β estradiolvalerat -eluting stent with that of the polymer-free rapamycin-eluting stent in patients with coronary artery disease. The ISAR stent is a rough surface stainless steel stent which allows coating without the need of polymer (PF ISAR stent) in the cath lab.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥50% de novo stenosis located in native coronary vessels.
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.

Exclusion Criteria:

* Target lesion located in the left main trunk or bypass graft.
* In-stent restenosis.
* Acute ST-elevation myocardial infarction.
* Cardiogenic shock.
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Known allergy to the study medications: aspirin, clopidogrel, rapamycin, estradiol, stainless steel.
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2005-03; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
in-stent late luminal loss | 6 months

SECONDARY OUTCOMES:
In-segment binary angiographic restenosis | 1 year
Need of target lesion revascularization | 1 year
Combined incidence of death or myocardial infarction | 1 year
Incidence of stent thrombosis. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schoemig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - 1. Medizinische Klinik, Klinikum rechts der Isar, München

REFERENCES:
- [Background] Sousa JE, Serruys PW, Costa MA. New frontiers in cardiology: drug-eluting stents: Part I. Circulation. 2003 May 6;107(17):2274-9. doi: 10.1161/01.CIR.0000069330.41022.90. No abstract available. PMID 12732594
- [Background] Babapulle MN, Joseph L, Belisle P, Brophy JM, Eisenberg MJ. A hierarchical Bayesian meta-analysis of randomised clinical trials of drug-eluting stents. Lancet. 2004 Aug 14-20;364(9434):583-91. doi: 10.1016/S0140-6736(04)16850-5. PMID 15313358
- [Background] Kastrati A, Dibra A, Eberle S, Mehilli J, Suarez de Lezo J, Goy JJ, Ulm K, Schomig A. Sirolimus-eluting stents vs paclitaxel-eluting stents in patients with coronary artery disease: meta-analysis of randomized trials. JAMA. 2005 Aug 17;294(7):819-25. doi: 10.1001/jama.294.7.819. PMID 16106007
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] McFadden EP, Stabile E, Regar E, Cheneau E, Ong AT, Kinnaird T, Suddath WO, Weissman NJ, Torguson R, Kent KM, Pichard AD, Satler LF, Waksman R, Serruys PW. Late thrombosis in drug-eluting coronary stents after discontinuation of antiplatelet therapy. Lancet. 2004 Oct 23-29;364(9444):1519-21. doi: 10.1016/S0140-6736(04)17275-9. PMID 15500897
- [Background] Wessely R, Kastrati A, Schomig A. Late restenosis in patients receiving a polymer-coated sirolimus-eluting stent. Ann Intern Med. 2005 Sep 6;143(5):392-4. doi: 10.7326/0003-4819-143-5-200509060-00119. Epub 2005 Aug 16. No abstract available. PMID 16106033
- [Background] Virmani R, Guagliumi G, Farb A, Musumeci G, Grieco N, Motta T, Mihalcsik L, Tespili M, Valsecchi O, Kolodgie FD. Localized hypersensitivity and late coronary thrombosis secondary to a sirolimus-eluting stent: should we be cautious? Circulation. 2004 Feb 17;109(6):701-5. doi: 10.1161/01.CIR.0000116202.41966.D4. Epub 2004 Jan 26. PMID 14744976
- [Background] Hausleiter J, Kastrati A, Wessely R, Dibra A, Mehilli J, Schratzenstaller T, Graf I, Renke-Gluszko M, Behnisch B, Dirschinger J, Wintermantel E, Schomig A; investigators of the individualizable durg-eluting Stent System to Abrogate Restenosis Project. Prevention of restenosis by a novel drug-eluting stent system with a dose-adjustable, polymer-free, on-site stent coating. Eur Heart J. 2005 Aug;26(15):1475-81. doi: 10.1093/eurheartj/ehi405. Epub 2005 Jun 23. PMID 15975990
- [Background] Mehilli J, Kastrati A, Wessely R, Dibra A, Hausleiter J, Jaschke B, Dirschinger J, Schomig A; Intracoronary Stenting and Angiographic Restenosis--Test Equivalence Between 2 Drug-Eluting Stents (ISAR-TEST) Trial Investigators. Randomized trial of a nonpolymer-based rapamycin-eluting stent versus a polymer-based paclitaxel-eluting stent for the reduction of late lumen loss. Circulation. 2006 Jan 17;113(2):273-9. doi: 10.1161/CIRCULATIONAHA.105.575977. Epub 2006 Jan 3. PMID 16391155
- [Background] Wessely R, Hausleiter J, Michaelis C, Jaschke B, Vogeser M, Milz S, Behnisch B, Schratzenstaller T, Renke-Gluszko M, Stover M, Wintermantel E, Kastrati A, Schomig A. Inhibition of neointima formation by a novel drug-eluting stent system that allows for dose-adjustable, multiple, and on-site stent coating. Arterioscler Thromb Vasc Biol. 2005 Apr;25(4):748-53. doi: 10.1161/01.ATV.0000157579.52566.ee. Epub 2005 Jan 27. PMID 15681298
- [Background] Dibra A, Kastrati A, Mehilli J, Pache J, Schuhlen H, von Beckerath N, Ulm K, Wessely R, Dirschinger J, Schomig A; ISAR-DIABETES Study Investigators. Paclitaxel-eluting or sirolimus-eluting stents to prevent restenosis in diabetic patients. N Engl J Med. 2005 Aug 18;353(7):663-70. doi: 10.1056/NEJMoa044372. Epub 2005 Aug 16. PMID 16105990
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Abizaid A, Albertal M, Costa MA, Abizaid AS, Staico R, Feres F, Mattos LA, Sousa AG, Moses J, Kipshidize N, Roubin GS, Mehran R, New G, Leon MB, Sousa JE. First human experience with the 17-beta-estradiol-eluting stent: the Estrogen And Stents To Eliminate Restenosis (EASTER) trial. J Am Coll Cardiol. 2004 Mar 17;43(6):1118-21. doi: 10.1016/j.jacc.2004.01.023. PMID 15028377
- [Result] Adriaenssens T, Mehilli J, Wessely R, Ndrepepa G, Seyfarth M, Wieczorek A, Blaich B, Iijima R, Pache J, Kastrati A, Schomig A. Does addition of estradiol improve the efficacy of a rapamycin-eluting stent? Results of the ISAR-PEACE randomized trial. J Am Coll Cardiol. 2007 Mar 27;49(12):1265-71. doi: 10.1016/j.jacc.2007.02.021. PMID 17394956